CLINICAL TRIAL: NCT01246492
Title: The Effect of Artificial Sweeteners on Blood Glucose Response
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Brain, Performance and Nutrition Research Centre, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 34AK1
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Taste Receptors; Nutrient Sensing; Intestinal Absorption; Blood Glucose; Appetite
MeSH Terms: interventions — Sweetening Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 45g glucose (Placebo Comparator): glucose water
  Interventions: Dietary Supplement: Artificial Sweeteners
- 45g glucose + 150mg aspartame (Active Comparator): glucose water aspartame
  Interventions: Dietary Supplement: Artificial Sweeteners
- 45g glucose + 20 mg saccharin (Active Comparator): glucose water saccharin
  Interventions: Dietary Supplement: Artificial Sweeteners
- 45g glucose + 85mg asculfame - K (Active Comparator): glucose water aseulfame- k
  Interventions: Dietary Supplement: Artificial Sweeteners

INTERVENTIONS:
Dietary Supplement: Artificial Sweeteners — A 400mL drink sweetened with 45g glucose and artificial sweetener will be consumed orally

SUMMARY:
The purpose of this study is to determine whether the presece of the artificial sweeteners aspartame, saccharin and asceulfame-k affect the blood glucose responses to an orally incested glucose solution.

DETAILED DESCRIPTION:
Sweet taste receptors, similar to those located on the lingual taste buds have been located along in the lining of the gut. Recent studies have demonstrated that activation of these sweetness taste receptors, either by sugars such as glucose, fructose, lactose, or artificial sweeteners such as saccharin and aspartame can influence the way nutrients, including glucose are absorbed from the gut into the bloodstream. Studies in animal models have shown that activation of the sweet taste receptors can increase the expression of the sodium-dependant glucose transporter 1 (SGLT1) and glucose transporter 2 (GLUT2) which transport glucose from the lumen into the bloodstream. Thus providing a potential mechanism by which glucose uptake can be regulated. Although artificial sweeteners stimulate the sweet taste receptors, they have little nutritive value, so that when they are consumed in the absence of any other nutrients there is little effect on blood glucose response. However, the effects of consuming artificial sweeteners in combination with sugars such as glucose is unclear. The purpose of this study is to investigate whether the addition of artificial sweeteners to an orally consumed glucose solution affects the rate at which the glucose appears in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Aged 18-45 years
* BMI (19-25 kg/m2)
* Weight stable in past 3 months

Exclusion Criteria:

* Smoking
* Females who are pregnant of breastfeeding
* Regular intake of emdication, other than females taking oral contraceptives
* Medical illness
* Gastrointestinal disorders
* Food allergies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Blood glucose response | 90 min
  Blood glucose will be determined at baseline and for 90 min following the consumption of the test drinks

SECONDARY OUTCOMES:
Subjective appetite | 90 min
  Subjective appetite ratings will be collected at baseline and for 90 min following the consumption of the test drinks

CONTACTS AND LOCATIONS:
Overall Officials: Nerys M Astbury, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance and Nutrition Research Centre- Northumbria University, Newcastle upon Tyne, United Kingdom